CLINICAL TRIAL: NCT06405789
Title: The Effect of Yoga on Mindfulness and Perceived Stress Level in Nursing Students
Brief Title: The Effect of Yoga on Mindfulness and Perceived Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özüm Erkin, Associate Professor, Izmir Democracy University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IDU-SBF-ÖE-01
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Stress
Keywords: yoga; mindfulness

STUDY DESIGN:
Intervention Model Description: A randomized controlled design with intervention and control groups.
Who Masked: Outcomes Assessor
Masking Description: A random allocation sequence was generated by an off-site statistician who was not involved in the participants' interventions. The statistician was given a class list of 69 people and asked to randomly assign them to groups A and B. The statistician did not know what A and B meant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The intervention group participated in 15 weeks of yoga/awareness activities led by the researcher. The yoga curriculum for the use of yoga in the classroom had been previously studied with nursing students and permission was obtained for its use in this study. The course content consists of 1.5 hours/per week (theoretical: 30 minutes; practical: 60 minutes) Each yoga session includes 5 minutes of breathing (pranayama) and warming up, 40 minutes of postures (asanas), 5 minutes of breathing (pranayama), 5 minutes of corpse pose (shavasana).In addition, to develop mindfulness, after the class, students were offered daily practices that enable a mindfulness-based approach to life events. The students participated in activities such as yoga practice, breathing and relaxation exercises, meditation practices with instructor notes and resources.
  Interventions: Other: yoga practice
- control (No Intervention): No intervention

INTERVENTIONS:
Other: yoga practice — The researcher has a yoga certificate before the study. The intervention group participated in 15 weeks of yoga/awareness activities led by the researcher. The yoga curriculum for the use of yoga in the classroom had been previously studied with nursing students and permission was obtained for its use in this study [11]. The course content consists of 1.5 hours/per week (theoretical: 30 minutes; practical: 60 minutes) Each yoga session includes 5 minutes of breathing (pranayama) and warming up, 40 minutes of postures (asanas), 5 minutes of breathing (pranayama), 5 minutes of corpse pose (shavasana).In addition, to develop mindfulness, after the class, students were offered daily practices that enable a mindfulness-based approach to life events. The students participated in activities such as yoga practice, breathing and relaxation exercises, meditation practices with instructor notes and resources.
  Arms: intervention

SUMMARY:
This study aimed to examine the effect of yoga on mindfulness and perceived stress levels in nursing students. A randomized controlled study was conducted in a nursing department in western Turkey between September 2019 and January 2020. The required institutional permission and ethics committee approval was received. The study participants were 56 nursing students with (intervention group (n:29), control group (n:27). The intervention group received the yoga program for 15 weeks delivered once a week. The control group did not practice yoga.

DETAILED DESCRIPTION:
This study aimed to examine the effect of yoga on mindfulness and perceived stress levels in nursing students in a parallel-group pretest-posttest randomized controlled study design. The required institutional permission and ethics committee approval was received.

The study was conducted in a nursing department in western Turkey between September 2019 and January 2020. The study consisted of 56 nursing students with (intervention group (n:29), control group (n:27). The intervention group received the yoga program for 15 weeks delivered once a week face to face. The control group did not practice yoga. The data were collected using "Personnel data form", "Mindful Attention Awareness Scale", "Perceived Stress Scale". The data were collected from the students using the online survey. For data analysis, descriptive statistics, paired sample t test, independent t, Pearson chi-square test were used. At the end of the study, the same yoga session was held with the students in the control group.

ELIGIBILITY:
Inclusion Criteria:

* being a first-year class nursing student
* older than 18 ages
* volunteering to participate
* giving consent

Exclusion Criteria:

* with a disability to practice yoga, hearing, and visual impairment
* unwillingness to continue participating in the study and school absenteeism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Mindful Attention Awareness Scale | 15 weeks
  The scale consists of fifteen items and consists of one dimension. The 6-point Likert-type scale has a rating scale of "1=almost always, 2=most of the time, 3=sometimes, 4=rarely, 5=very rarely, 6=almost never". While this scale provides a single total score, high scores indicate high levels of mindfulness
Perceived Stress Scale (PSS) | 15 weeks
  The PSS, which consists of a total of 10 items, was developed to measure the extent to which certain situations in a person's life are perceived as stressful. Participants rated each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". While The scores of the PSS-10 range from 0 to 40 and from 0 to 16. A high score indicates an increased perception of stress

CONTACTS AND LOCATIONS:
Overall Officials: özüm erkin, Ph.D, Principal Investigator — İzmir Democracy University
Locations (1):
- İzmir Democracy University, Izmir, Ege Bölgesi, Turkey (Türkiye)